CLINICAL TRIAL: NCT04436016
Title: Effect of Heart Rate Control With Ivabradine on Myocardial Injury After Non-cardiac Surgery: a Single Center, Randomized Controlled, Double-blind Feasibility Pilot Trial
Brief Title: PeRiOperaTivE CardioproTection With Ivabradine in Non-cardiac Surgery
Acronym: PROTECTIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Bernardo Bollen Pinto, MD PhD, Senior Registrar and Research Fellow, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PROTECTIN Pilot; SNCTP000003728 (Registry Identifier: Swiss Federal Office of Public Health's portal for human research)
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Myocardial Injury; Myocardial Ischemia
Keywords: ivabradine; heart rate; pilot study; myocardial injury after non-cardiac surgery; perioperative myocardial injury; feasibility study; perioperative medicine
MeSH Terms: conditions — Myocardial Ischemia | interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: Single center, randomized, placebo-controlled, double-blind, parallel group, feasibility pilot trial.
  Patients will be randomized to receive ivabradine or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine (Experimental): Ivabradine will be administered in an individualized regimen adapted to the subject's heart rate at each visit in a dosage ranging from 0-7.5mg twice daily (morning and evening) from the morning of surgery until post-operative day 2, as follows:
  * If heart rate is ≥101 bpm: capsule D (Ivabradine 7.5 mg);
  * If heart rate is 86-100 bpm: capsule C (Ivabradine 5 mg);
  * If HR is 71-85 bpm: capsule B (Ivabradine 2.5 mg);
  * If HR ≤ 70 bpm or the patient received rescue treatment for bradycardia (eg.atropine) after the previous dose: capsule A (placebo).
  Interventions: Drug: Ivabradine; Drug: Placebo
- Placebo (Placebo Comparator): Placebo will be administered twice daily (morning and evening) from the morning of surgery until post-operative day 2, as follows:
  * If heart rate is ≥101 bpm: capsule D (Placebo)
  * If heart rate is 86-100 bpm: capsule C (Placebo)
  * If HR is 71-85 bpm: capsule B (Placebo)
  * If HR ≤ 70 bpm or the patient received rescue treatment for bradycardia (eg.atropine) after the previous dose: capsule A (Placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Ivabradine pills will be crushed and encapsulated for adequate dosing (0, 2.5mg, 5mg or 7.5 mg) and blinding.
  Other Names: Procoralan
  Arms: Ivabradine
Drug: Placebo — Mannitol will be encapsulated for adequate blinding.

SUMMARY:
Perioperative myocardial injury (PMI) after non-cardiac surgery (NCS), i.e. the elevation of postoperative troponin, occurs in nearly 20% of patients older than 45 years undergoing NCS and is independently and strongly associated with post-operative mortality (30-day mortality up to 10%). With over 300 million surgical interventions every year worldwide, PMI has a high clinical relevance on the health of the population.

Heart rate (HR) is an independent and modifiable risk factor for PMI and death after non-cardiac surgery. Numerous studies showed that beta-blockers decrease myocardial ischemia after surgery in a heart-rate dependent manner, but this beneficial effect is surpassed by an increased incidence of perioperative hypotension and death. Currently, no single intervention is available to decrease the risk of perioperative cardiac complications. Ivabradine (IVA) is a negative chronotropic agent without significant effects on contractility or vascular tone and has been shown to improve outcomes in the setting of chronic and acute heart diseases.

Rationale for pilot feasibility trial: the planned definitive large trial is a multicenter trial to investigate the efficacy of ivabradine to decrease perioperative myocardial injury. The intervention planned is complex and demands important resources. The investigators designed this pilot study to inform on the feasibility of the definitive large trial. This pilot study will also provide additional information that could help investigators improve the definitive large trial regarding recruitment, refinements to the study protocol and improving the participant's experience.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature of patient; AND
* Undergoing intermediate or high-risk non-cardiac surgery (as defined in European Society of Anaesthesiology guidelines) AND;
* One of the following:

  o≥ 75 years old OR; o≥ 45 years old AND at least 1 risk factors independently associated with perioperative myocardial injury (history of coronary artery disease, chronic heart failure, peripheral artery disease, ischemic stroke, hypertension, diabetes mellitus, chronic kidney disease).

Exclusion Criteria:

* Inability to provide informed consent;
* History of hypersensitivity or allergy to ivabradine;
* Emergency surgery (to be done within 24h of diagnosis);
* Shock or acute decompensated heart failure at trial inclusion;
* Low cardiac output syndrome;
* Arrhythmia:

  * Atrial fibrillation or flutter;
  * AV-block of 3rd degree;
  * Sick sinus syndrome;
  * Sino-atrial block;
* Pacemaker dependency;
* Unstable angina;
* Acute myocardial infarction in the 3 months preceding the trial;
* Stroke in the 3 months preceding the trial;
* Cirrhosis Child B and C;
* Renal failure with a Estimated Glomerular filtration rate ≤ 15 ml/min/1.73m2;
* Treatment with a strong cytochrome P450 3A4 inhibitors such as azole antifungals (ketoconazole, itraconazole), macrolide antibiotics (clarithromycin, erythromycin; josamycin, telithromycin), HIV protease inhibitors (nelfinavir, ritonavir) and nefazodone;
* Treatment with verapamil or diltiazem which are moderate CYP3A4 inhibitors and PGP inducers with heart rate reducing properties;
* Women who are pregnant or breast feeding;
* Childbearing potential (Of note, woman with history of hysterectomy, surgical sterilization or menopause for longer than 2 years are not considered with childbearing potential, independent of their age);
* Participation in another study with investigational drug within the 30 days preceding and during the present study;
* Previous enrolment into the current study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Appropriate dosage rate | From the morning (6-9 am) of the day of surgery of the first study participant to the evening of the second post-operative day of the last study participant (up to 1 year from first randomization).
  Number of correct dosages administered according to the patient's heart rate at each study visit divided by the total dosages administrated
Blinding success rate | From the morning (6-9 am) of the day of surgery of the first study participant to the evening of the second post-operative day of the last study participant (up to 1 year from first randomization).
  Number of times blinding code was broken divided by the total dosages administrated

SECONDARY OUTCOMES:
Recruitment rate | Up to one year from the date participant screening begins.
  Total number of eligible participants approached, the number recruited and randomised divided by the number of months that the trial recruited for
Participant satisfaction regarding information about the study, informed consent, recruitment procedures and study participation | Screening, morning of the day surgery pre-operatively and post-operative days 1, 2 and 3.
  Qualitative research methods (shadowing and semi-structured interviews)
Perioperative myocardial injury | Day of surgery pre-operatively (between 6-9 am) and post-operatively (between 6-9 pm or within 1h after surgery if surgery ends after 9pm) and morning (between 6-9 am) of post-operative days 1, 2, 3 and day of hospital discharge.
  Variance of high-sensitive cardiac troponin T (ng/L)
Heart rate | Day of surgery pre-operatively (between 6-9 am) and post-operatively (between 6-9 pm or within 1h after surgery if surgery ends after 9pm) and morning (between 6-9 am) of post-operative days 1, 2, 3 and day of hospital discharge.
  Variance of resting heart rate
Ivabradine dosage | Day of surgery pre-operatively (between 6-9 am) and morning (between 6-9 am) of post-operative days 1 and 2.
  Variance
Quality of Recovery | Morning (between 6-9 am) of post-operative days 1, 3 and at day of hospital discharge.
  Variance of Quality of Recovery assessed with Quality of Recovery-15 scale (range from 0 to 150, with higher scores indicating a better outcome)
Difficulty in following study protocol and administrating study drug | Morning (between 6 and 9 am) and evening (between 6 and 9 pm) of day of sugery and post-operative days 1 and 2.
  4-point Likert scale (Study personnel will be asked "The decision to administer the study drug according to the patient's heart rate was straightforward". Answers range from Strongly agree, Agree, Disagree to Strongly disagree)

OTHER OUTCOMES:
Bradycardia | From the morning of the day of surgery when the first study intervention (between 6-9am) is adminitstered until post-operative day 3 in the morning (between 6-9am).
  Number of patients with those with a heart rate <50 or requiring an intervention to increase heart rate as atropine
Atrial fibrilation | From the morning of the day of surgery when the first study intervention (between 6-9am) is adminitstered until post-operative day 3 in the morning (between 6-9am).
  Number of patients with atrial fibrilation
Phosphenes | From the morning of the day of surgery when the first study intervention (between 6-9am) is adminitstered until post-operative day 3 in the morning (between 6-9am).
  Number of patients with phosphenes
NT-proBNP | Day of surgery post-operatively (between 6-9 pm) and morning (between 6-9 am) of post-operative days 1, 2 and 3.
  Variance of NT-proBNP (pg/L)
Cardiac output (CO) | Day of surgery post-operatively (between 6-9 pm) and morning (between 6-9 am) and evening (betwee 6-9pm) of post-operative days 1, 2 and 3.
  Variance of CO measured with the ICON monitor (L/min)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Bollen Pinto, MD PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puelacher C, Lurati Buse G, Seeberger D, Sazgary L, Marbot S, Lampart A, Espinola J, Kindler C, Hammerer A, Seeberger E, Strebel I, Wildi K, Twerenbold R, du Fay de Lavallaz J, Steiner L, Gurke L, Breidthardt T, Rentsch K, Buser A, Gualandro DM, Osswald S, Mueller C; BASEL-PMI Investigators. Perioperative Myocardial Injury After Noncardiac Surgery: Incidence, Mortality, and Characterization. Circulation. 2018 Mar 20;137(12):1221-1232. doi: 10.1161/CIRCULATIONAHA.117.030114. Epub 2017 Dec 4. PMID 29203498
- [Background] Duceppe E, Parlow J, MacDonald P, Lyons K, McMullen M, Srinathan S, Graham M, Tandon V, Styles K, Bessissow A, Sessler DI, Bryson G, Devereaux PJ. Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment and Management for Patients Who Undergo Noncardiac Surgery. Can J Cardiol. 2017 Jan;33(1):17-32. doi: 10.1016/j.cjca.2016.09.008. Epub 2016 Oct 4. PMID 27865641
- [Background] Chen A, Elia N, Dunaiceva J, Rudiger A, Walder B, Bollen Pinto B. Effect of ivabradine on major adverse cardiovascular events and mortality in critically ill patients: a systematic review and meta-analyses of randomised controlled trials with trial sequential analyses. Br J Anaesth. 2020 Jun;124(6):726-738. doi: 10.1016/j.bja.2020.01.027. Epub 2020 Mar 6. PMID 32147100
- [Background] Abbott TEF, Pearse RM, Archbold RA, Ahmad T, Niebrzegowska E, Wragg A, Rodseth RN, Devereaux PJ, Ackland GL. A Prospective International Multicentre Cohort Study of Intraoperative Heart Rate and Systolic Blood Pressure and Myocardial Injury After Noncardiac Surgery: Results of the VISION Study. Anesth Analg. 2018 Jun;126(6):1936-1945. doi: 10.1213/ANE.0000000000002560. PMID 29077608
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Derived] White MJ, Zaccaria I, Ennahdi-Elidrissi F, Putzu A, Dimassi S, Luise S, Diaper J, Mulin S, Baudat AD, Gil-Wey B, Elia N, Walder B, Bollen Pinto B. Personalised perioperative dosing of ivabradine in noncardiac surgery: a single-centre, randomised, placebo-controlled, double-blind feasibility pilot trial. Br J Anaesth. 2024 Oct;133(4):738-747. doi: 10.1016/j.bja.2024.05.020. Epub 2024 Jul 2. PMID 38960832